CLINICAL TRIAL: NCT01575587
Title: A Single-Dose, Open-Label, Randomized, 4-Way Crossover Study to Assess the Effect of Timing of Food Intake on the Pharmacokinetics of Abiraterone Following Single-Dose Administration of Abiraterone Acetate Tablets in Healthy Caucasian and Japanese Male Subjects
Brief Title: A Study to Assess the Effect of Timing of Food Intake on the Pharmacokinetics of Abiraterone Following Single-Dose Administration of Abiraterone Acetate Tablets in Healthy Caucasian and Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100737; 212082PCR1005 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-01-19; First posted 2012-04-11 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Pharmacology
Keywords: Pharmacology; Pharmacokinetics; Pharmacodynamics; Abiraterone acetate; Food intake; Caucasion; Japanese; Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: Abiraterone: Treatment A
- Treatment B (Experimental)
  Interventions: Drug: Abiraterone: Treatment B
- Treatment C (Experimental)
  Interventions: Drug: Abiraterone: Treatment C
- Treatment D (Experimental)
  Interventions: Drug: Abiraterone: Treatment D

INTERVENTIONS:
Drug: Abiraterone: Treatment A — 1000 mg abiraterone acetate administered in the fasting state
  Arms: Treatment A
Drug: Abiraterone: Treatment B — Standardized meal administered 1 hour after the 1000 mg abiraterone acetate dose
  Arms: Treatment B
Drug: Abiraterone: Treatment C — Standardized meal administered 2 hours before the 1000 mg abiraterone acetate dose
  Arms: Treatment C
Drug: Abiraterone: Treatment D — Standardized meal administered 2 hours before and 2 hours after the 1000 mg abiraterone acetate dose
  Arms: Treatment D

SUMMARY:
The purpose of this study is to evaluate the effect of timing of food intake on systemic abiraterone exposure observed in healthy adult Japanese and Caucasian men.

DETAILED DESCRIPTION:
This is a randomized (individuals will be assigned by chance to study treatments), open-label (individuals will know the identity of study treatments), single dose, 4-way crossover study of abiraterone acetate in approximately 48 healthy adult Japanese and Caucasian men. For the crossover design, the treatment sequences are defined as follows: 1 - ADBC, 2 - BACD, 3 - CBDA, and 4 - DCAB; where Treatment A = abiraterone acetate administered in the fasted state, Treatment B = standardized meal administered 1 hour after abiraterone acetate dose, Treatment C = standardized meal administered 2 hours after abiraterone acetate dose, and Treatment D = standardized meal administered 2 hours before and 2 hours after abiraterone acetate dose. This study will consist of a screening period followed by four open-label treatment periods separated by a washout period of at least 14 days between dosing. Eligible participants will be randomly assigned on Day 1 to 1 of 4 treatment sequences that differ with regard to timing of food intake before and/or after dosing with a single dose of 1000 mg of abiraterone acetate. Serial pharmacokinetic (study of what the body does to a drug) samples will be collected during the open-label treatment phase as detailed in the protocol. Safety will be monitored throughout the study. End-of-study assessments will be performed on Day 4 of Period 4 or upon early withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian and Japanese male individuals.
* Body mass index between 18 and 30 kg/m2.
* Body weight >=50 kg.
* A normal 12-lead electrocardiogram.

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results.
* Presence of sexual dysfunction (abnormal libido, erectile dysfunction, etc.) or any medical condition that would affect sexual function.
* History of alcohol consumption of more than 4 drinks daily within 1 year prior to screening and unwillingness to abstain from alcohol-containing food or beverages from within 24 hours before Day-1 through study completion.
* History of, or a reason to believe a participant has a history of drug or alcohol abuse within the past 5 years.
* Positive test for human immunodeficiency virus 1 and 2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
* History of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or participant's verbal report.

Ages: 25 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Changes in mean plasma concentrations of abiraterone | Up to Day 4, treatment period 4

SECONDARY OUTCOMES:
Mean plasma concentrations of abiraterone | Up to Day 4, treatment period 4
Maximum plasma concentration of abiraterone | Up to Day 4, treatment period 4
Time to reach the maximum plasma concentration of abiraterone | Up to Day 4, treatment period 4
Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentration of abiraterone | Up to Day 4, treatment period 4
Area under the plasma concentration-time curve from time 0 to infinite time of abiraterone | Up to Day 4, treatment period 4
Elimination half-life associated with the terminal slope of the semilogarithmic drug concentration-time curve of abiraterone | Up to Day 4, treatment period 4
First-order rate constant associated with the terminal portion of the curve of abiraterone | Up to Day 4, treatment period 4
Time to last quantifiable plasma concentration of abiraterone | Up to Day 4, treatment period 4
Percentage of area under the plasma concentration-time curve from time 0 to infinite time obtained by extrapolation of abiraterone | Up to Day 4, treatment period 4
The number of participants affected by an adverse event | Up to the end of the study (4 days after final dose of study drug) or early withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States

REFERENCES:
- [Derived] Inoue K, Shishido A, Vaccaro N, Jiao J, Stieltjes H, Bernard A, Yu M, Chien C. Pharmacokinetics of abiraterone in healthy Japanese men: dose-proportionality and effect of food timing. Cancer Chemother Pharmacol. 2015 Jan;75(1):49-58. doi: 10.1007/s00280-014-2616-4. Epub 2014 Oct 25. PMID 25344090